CLINICAL TRIAL: NCT00439920
Title: GIMEMA LAL 0496: High-dose Anthracycline in the Induction Regimen for the Treatment of Adult Acute Lymphoblastic Leukemia. A Prospective Multicentric GIMEMA Trial.
Brief Title: GIMEMA LAL 0496: High-dose Anthracycline in the Induction Regimen for the Treatment of Adult ALL.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL0496
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Anthracyclines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-dose anthracycline (Experimental)
  Interventions: Drug: High-dose anthracycline

INTERVENTIONS:
Drug: High-dose anthracycline

SUMMARY:
The present study aims at verifying the state of the art in what this illness concerns and at organizing a centralized samples analysis.

DETAILED DESCRIPTION:
The present trial is a prospective multicentric GIMEMA study, in which adult ALL patients are extensively analyzed at diagnosis by a multiparametric approach including CC and molecular analysis for the following gene rearrangements: BCR-ABL, MLL-AF4, E2A-PBX1, TEL-AML1, MLL, p15 and p16 deletion in order to give place to a carefully characterization of the genetic lesions occurring in adult ALL and to evaluate their prognostic significance in a large cohort of patients homogeneously treated.

This study requires a central handling and analysis of bone marrow (BM) or peripheral blood samples at presentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-60
* Diagnosed with previously untreated T-ALL and B-ALL

Exclusion Criteria:

* previously treated ALL patients
* L3 B-ALL

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1996-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete response
  Patients are followed-up for response till death

SECONDARY OUTCOMES:
Number of patients that reach disease-free-survival
  Patients are followed-up for response till death

CONTACTS AND LOCATIONS:
Overall Officials: Franco Mandelli, Prof., Principal Investigator — Università degli Studi di Roma "La Sapienza"

REFERENCES:
- [Derived] Piciocchi A, Messina M, Elia L, Vitale A, Soddu S, Testi AM, Chiaretti S, Mancini M, Albano F, Spadano A, Krampera M, Bonifacio M, Cairoli R, Vetro C, Colella F, Ferrara F, Cimino G, Bassan R, Fazi P, Vignetti M. Prognostic impact of KMT2A-AFF1-positivity in 926 BCR-ABL1-negative B-lineage acute lymphoblastic leukemia patients treated in GIMEMA clinical trials since 1996. Am J Hematol. 2021 Sep 1;96(9):E334-E338. doi: 10.1002/ajh.26253. Epub 2021 Jun 9. No abstract available. PMID 34048072